CLINICAL TRIAL: NCT05595655
Title: Tailored Intervention for Self-Care Promotion in Patients With Heart Failure: Protocol for a Randomized Controlled Trial to Test the Efficacy of Motivational Interviewing on Self-care
Brief Title: Randomized Controlled Trial to Test the Efficacy of Motivational Interviewing on Self-care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale di Lodi (Other)
Responsible Party: Principal Investigator, Greta Ghizzardi, Principal Investigator, Azienda Socio Sanitaria Territoriale di Lodi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Asstlodi-Oct22
Record Dates: First submitted 2022-10-20; First posted 2022-10-27 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure
Keywords: heart failure; motivational interviewing; self-care
MeSH Terms: conditions — Heart Failure | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): The dyads will receive traditional educational treatment only and will complete the questionnaires after 3, 6, 9 and 12 months follow-up post-intervention. Enrolled dyads will be monitored by the research team responsible for recruitment and follow-up.
- First interventional arm (Other): MI intervention will be administered to patients only and caregivers will receive standard education. The intervention will last approximately 30 minutes. Thereafter, the nurse who performed the MI will contact the patients over the phone 3 times during the first 2 months after MI, to strengthen the intervention. Then, the intervention will be employed again after 3, 6, 9 and 12 months from enrolment. After each MI session, both patients and caregivers will be asked to complete the questionnaires of follow-up post-intervention
  Interventions: Behavioral: Motivational Interviewing
- Second interventional arm (Experimental): MI intervention will be administered both to patients and caregivers. The intervention will be administered to the dyad in one session and patients and their caregivers will receive the reinforcing educational treatment calibrated on the specific lacking areas of patients' self-care behaviours. After each MI session, both patients and caregivers will be asked to complete the questionnaires of follow-up post-intervention.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interviewing (MI) is a directive client-centred counselling approach for eliciting behavioral change by helping people to explore and resolve ambivalence. MI considers several critical factors to improving self-care in patients with HF and is based on brief interventions, which are feasible in several healthcare settings.
  Arms: First interventional arm; Second interventional arm

SUMMARY:
Introduction: Heart failure (HF) is characterized by an increasing prevalence and burden, representing a public health problem and a major cause of morbidity and mortality. Self-care is a cornerstone approach for optimizing therapy for patients with HF; patients play a key role in the management of their condition, given that several negative health outcomes might be avoided with effective self-care. Motivational interviewing (MI) has been described by the literature as highly favorable for treating chronic diseases, with promising results supporting its efficacy in enhancing self-care. Moreover, caregivers' availability constitutes a fundamental supporting factor among the strategies to improve self-care behaviors in people with HF.

Methods and analysis: This study protocol designed a prospective, parallel-arm, open-label, three-arm, controlled trial for purposing the aims to test the efficacy of a structured program including scheduled MI interventions in improving self-care behaviors among patients with HF at 3, 6, 9, and 12 months from the enrolment. Secondary aims comprehend the corroboration of the superiority of caregivers' participation to the structured program including scheduled MI interventions over the program administrated only to individual patients in enhancing self-care behaviors and other outcomes. Analyses will be performed within the framework of intention-to-treat (ITT). Comparisons between groups will be based on an alpha = 5% and two-tailed null hypotheses. In the case of missingness, analyzing the extent of the missingness and identifying underlying mechanisms and patterns will guide imputation methods.

Ethics and dissemination: The study protocol and template consent forms have been reviewed and approved by the Ethical Committee of San Raffaele Hospital (approval #74/INT). Also, the study protocol has been registered at ClinicalTrials.gov (Identifier: …….). Patients and caregivers will have to sign the informed consent forms before the randomisation. Patients and caregivers may leave the study at any time. The withdrawal from the study will not imply any prejudice, as fully documented and explained in the informed consent. Considering the open-access publication, the full protocol will be available freely.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* diagnosis of HF with New York Heart Association (NYHA) Class II-IV;
* no acute coronary events within three months;
* consent to participate in the study;
* score ≤ 2 to at least two items of the Self-Care of Heart Failure Index 6.2 - SCHFI 6.2 at baseline;
* score on Six Item Screener > 4;
* living at home;
* understanding of spoken and written Italian.

Exclusion Criteria:

* severe cognitive impairment (score 0-4 on the Six-item Screener);
* acute coronary events that occurred within three months;
* living in nursing homes or residential settings;
* caregivers unwilling to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Changes will be assessed in the Level of self-care maintenance - Self-Care of Heart Failure Index 6.2 | 3, 6, 9, and 12 months from the enrollment
  self-care behavior consisting in keeping the disease stable

SECONDARY OUTCOMES:
Changes will be assessed in the Level of caregivers' involvement - Caregiver Contribution to Self-care of Heart Failure Index (CC-SCHFI) | 3, 6, 9, and 12 months from the enrollment
  superiority of the caregivers' participation to the structured program including scheduled MI interventions over the program administrated only to individual patients in enhancing self-care behaviors
Changes will be assessed in the Level of patient's ability to feel the symptoms of HF - Heart Failure Somatic Perception Scale (HFSPS) | 3, 6, 9, and 12 months from the enrollment
  patient's ability perceive the symptoms of HF
Changes will be assessed in the Level of cognitive impairment- Six Item Screener | 3, 6, 9, and 12 months from the enrollment
  patients' cognitive impairment
Changes will be assessed in the Level of physical function, symptoms, social function, self-efficacy, and quality of life (QoL) - Kansas City Cardiomyopathy Questionnaire (KCCQ) | 3, 6, 9, and 12 months from the enrollment
  HF-specific QoL
Changes will be assessed in the Level of feeling of intimacy and positive relationship between patient and caregiver -Mutuality Scale (MS) | 3, 6, 9, and 12 months from the enrollment
  feeling of intimacy and positive relationship between patient and caregiver
Changes will be assessed in the Level of physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health - SF-12 | 3, 6, 9, and 12 months from the enrollment
  generic health-related QoL
Changes will be assessed in the Level of presence of significant sleep disturbance experienced in the month before the assessment - Pittsburgh Sleep Quality Index (PSQI) | 3, 6, 9, and 12 months from the enrollment
  sleep quality
Changes will be assessed in the Level of depression and anxiety - Hospital Anxiety and Depression Scale (HADS) | 3, 6, 9, and 12 months from the enrollment
  depression and anxiety
Changes will be assessed in the Level of cognitive impairment - Montreal Cognitive Assessment (MoCA) | 3, 6, 9, and 12 months from the enrollment
  mild cognitive impairment
Changes will be assessed in the Number of comorbidities - Charlson Comorbidity Index (CCI) | 3, 6, 9, and 12 months from the enrollment
  comorbidities
Changes will be assessed in the Level of caregiver contribution to self-care - Caregiver Contribution to Self-care of Heart Failure Index (CC-SCHFI) | 3, 6, 9, and 12 months from the enrollment
  caregiver contribution to self-care in patients with HF
Changes will be assessed in the Level of caregiver Preparedness - Caregiver Preparedness Scale (CPS) | 3, 6, 9, and 12 months from the enrollment
  Caregiver Preparedness to care
Changes will be assessed in the Level of social support - Multidimensional Scale of Perceived Social Support (MSPSS) | 3, 6, 9, and 12 months from the enrollment
  level of social support perceived by HF patients in managing the disease

CONTACTS AND LOCATIONS:
Overall Officials: Federica Dellafiore, Principal Investigator — Università degli Studi di Pavia
Locations (1):
- Cardiology, Lodi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
raw data sharing

REFERENCES:
- [Derived] Dellafiore F, Ghizzardi G, Vellone E, Magon A, Conte G, Baroni I, De Angeli G, Vangone I, Russo S, Arrigoni C, Caruso R. Motivational Interviewing for Enhancing Self-care in Patients With Heart Failure: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 28;12:e44629. doi: 10.2196/44629. PMID 36976630